CLINICAL TRIAL: NCT03483779
Title: A Series of N-of-1 Trials of Comparing Ginkgo Biloba Pills and Placebo in the Treatment of Coronary Heart Disease With Impaired Glucose Regulation
Brief Title: Comparing Ginkgo Biloba Pills and Placebo in the Treatment of Coronary Heart Disease With Impaired Glucose Regulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Wanbangde Pharmaceutical Group Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YXY20180226
Record Dates: First submitted 2018-03-25; First posted 2018-03-30 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-02

CONDITIONS: Randomized Controlled Trial; Ginkgo Biloba Extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group:Ginkgo biloba pills (Experimental): Five Ginkgo biloba pills a time and three times a day. One treatment period including 8 weeks.
  Interventions: Drug: Ginkgo biloba pills
- Control group:placebo pills (Placebo Comparator): Five placebo pills a time and three times a day. One treatment period including 8 weeks.
  Interventions: Drug: placebo pills

INTERVENTIONS:
Drug: Ginkgo biloba pills — Each N-of-1 trial will consist of 6 treatment periods, of which 2 treatment periods are in one group, including 8 weeks of placebo treatment and 8 weeks of ginkgo biloba pills.
  Arms: Experimental group:Ginkgo biloba pills
Drug: placebo pills — Each N-of-1 trial will consist of 6 treatment periods, of which 2 treatment periods are in one group, including 8 weeks of placebo treatment and 8 weeks of ginkgo biloba pills.
  Arms: Control group:placebo pills

SUMMARY:
Background

Coronary heart disease has become a serious challenge to China with its high prevalence and mortality. The impaired glucose regulation is prevalent in patients with cardiovascular disease. However, there are few drugs that interfere early with impaired glucose regulation. Ginkgo biloba extract is not only a commonly used drug for cardiovascular diseases, but also has a significant effect in reducing blood sugar. Therefore, this study used a single case randomized controlled trial to explore the efficacy of Ginkgo biloba pills in the treatment of coronary heart disease patients with impaired glucose regulation.

Methods

This is a randomized, double-blind, placebo-controlled, three-period crossover trial for a single subject.A total of 12 subjects will be recruited in this trial. The trial is divided into three cycles, one cycle has two treatment periods. Ginkgo biloba pills and placebo will be randomized during the treatment period. The test period will be lasted 58 weeks and subjects will take 48 weeks. Subjects will be selected by the researcher strictly in accordance with the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. male and female patients with clear history of previous myocardial infarction or history of percutaneous coronary intervention（PCI） or history of coronary artery bypass grafting(CABG) (at least 3 months or more),or who have coronary angiography or coronary CT angiography（CTA） results suggested at least one coronary artery stenosis and lumen stenosis ≥50%,
2. in line with the criteria for stable angina, and the number of episodes of angina pectoris ≥ 2 times per week,
3. comply with the diagnostic criteria of blood stasis syndrome of coronary heart disease（CHD）,
4. comply with the 2016 Diabetes Association (ADA) published criteria for impaired diagnosis of glucose regulation，
5. aged between 18 and 75 years，
6. participants voluntarily participated in this study, signed informed consent and had good compliance.

Exclusion Criteria:

1. with congenital or rheumatic heart disease or severe cardiopulmonary insufficiency (grade 3 and 4 of cardiac function),or uncontrolled severe arrhythmias (including ventricular tachycardia, supraventricular tachycardia),or not controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure≥ 100 mmHg),
2. with cerebrovascular disease,or with severe liver and kidney dysfunction, or with endocrine, urinary, blood system and other serious primary diseases,
3. within 4 weeks, there was history of major organ surgery such as head, chest or abdomen or bleeding tendency,
4. those who have taken hypoglycaemic agents or glucocorticoids, thiazide diuretics and other drugs that affect blood sugar levels within 3 months,
5. people with diseases affecting blood glucose metabolism, such as thyroid glands and adrenal diseases, or those with previous history of the aforementioned diseases,
6. allergies or persons allergic to known ingredients of the study drug,
7. pregnancy and lactation women or those with a pregnancy plan,
8. subjects who participated in other clinical trials in the last 3 months,
9. researchers consider that subjects should not participate in clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-04-25 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
fasting plasma glucose (FPG) | 8 weeks
  changes in blood glucose
postprandial 2h blood glucose (2hPG) | 8 weeks
  changes in blood glucose
Seattle Angina Questionnaire | 8 weeks
  Questionnaires will be completed (SAQ - Seattle Angina Questionnaire) at the end of each treatment period.
  The Seattle Angina Questionnaire (SAQ) is a self-administered, 19-item questionnaire, a cardiac disease-related quality-of-life measure. The SAQ is well validated and sensitive to clinical changes. It has five subscales: physical limitation, angina stability, angina frequency, treatment satisfaction, and quality of life. The possible range of scores for each of the five subscales is 0 to 100, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Symptoms of angina pectoris | 8 weeks
  Symptoms of angina pectoris, including frequency, duration, attack severity, and the doses of nitroglycerin were recorded, and an angina pectoris symptom score will be calculated. The effect index is determined according to the following formula:
  Effect index (n) = [(symptom score before treatment - symptom score after treatment) / symptom score before treatment] × 100%.
  A value of n ≥ 70% suggested a significant effect; 70% >n ≥ 30% suggested an effect; 30% >n ≥ 0 suggested no effect; n < 0 suggested a worsening effect.
C-reactive protein | 8 weeks

OTHER OUTCOMES:
HbA1c | 8 weeks
fasting insulin | 8 weeks
lipids | 8 weeks
main adverse cardiovascular and cerebrovascular events(MACCE) | 58 weeks
  incidence of composite endpoints of major adverse cardiovascular and cerebrovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Rui Gao, PhD, Study Chair — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun M, Chai L, Lu F, Zhao Y, Li Q, Cui B, Gao R, Liu Y. Efficacy and Safety of Ginkgo Biloba Pills for Coronary Heart Disease with Impaired Glucose Regulation: Study Protocol for a Series of N-of-1 Randomized, Double-Blind, Placebo-Controlled Trials. Evid Based Complement Alternat Med. 2018 Oct 14;2018:7571629. doi: 10.1155/2018/7571629. eCollection 2018. PMID 30405743